CLINICAL TRIAL: NCT04613102
Title: The Efficacy and Safety of 3% Cannabidiol (CBD) Cream in Patients With Epidermolysis Bullosa: A Phase II/III Trial
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study protocol should to be updated (major updates), following the second Health Canada review /requests. The study has been withdrawn form the REB review and will not be performed at SickKids.
Sponsor: Elena Pope (Other)
Collaborators: Avicanna Inc (Industry)
Responsible Party: Sponsor-Investigator, Elena Pope, Dermatology section head, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1000062062
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Epidermolysis Bullosa; Pain; Itch
MeSH Terms: conditions — Epidermolysis Bullosa; Pain; Pruritus

STUDY DESIGN:
Intervention Model Description: Phase 2 of the study is open label . Phase 3 study participants will be his own control: they will be treated by the active medication ( AVCN583601) and placebo simultaneously during full study treatment period, applying thestudy cream from two different jars to two different body sides ( left/right).
Who Masked: Participant, Investigator
Masking Description: Only phase 3 of the clinical trial is going to be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- interventional arm, phase 2 (Experimental): All participant of phase 2 will receive CBD cream for their chronic wound treatment.
  This is an open-label part of the study.
  Interventions: Drug: AVCN583601 (3% Cannabidiol cream)
- Interventional arm, phase 3 (Experimental): Each participants of the phase 3 will receive the active study medication (AVCN583601) during the entire study treatment period on the one of his body sides, and placebo cream - on the other body side simultaneously (left/right). So, each participant will be his own control.
  The research support pharmacy will randomize, which side of the body participant should apply CBD cream on, and provide two jars with the study medications, labeled accordingly ( Left /Right).
  Interventions: Drug: AVCN583601 (3% Cannabidiol cream)

INTERVENTIONS:
Drug: AVCN583601 (3% Cannabidiol cream) — Topical application twice daily for 4 weeks (phase 2) and for 8 weeks (phase 3).
  Other Names: Cannabidiol cream

SUMMARY:
Epidermolysis bullosa (EB) is rare, devastating, and currently incurable genetic blistering disorders characterized by fragility of skin and mucosal membranes. Therapeutic options for EB are limited. Acute and chronic wounds cause pain, itching and infection, altering quality of life and impair wound healing. In absence of a cure, wound care is paramount to alleviate suffering.

Anecdotal experience suggest that CBD application alleviates the pain and itching and improves wound healing by controlling the inflammatory process. We propose to undertake a phase II/III study exploring the safety, tolerability and efficacy of topical application of 3% Cannabidiol cream (CBD) on acute and chronic wounds affecting patients with EB.

We are doing this trial to determine safety and tolerability of topical CBD cream in a cohort of RDEB patients with chronic wounds (phase II trial), and to evaluate the efficacy and safety of CBD cream in EB with acute and chronic wounds in promoting wound healing, decrease blister formation, pain, itching and improve overall quality of life (phase III trial)

DETAILED DESCRIPTION:
Phase II is an open-label part of the study. We are planning to enroll in this phase 10 patients, diagnosed with Epidermolysis Bullosa with chronic wounds , and treat them with topical application of 3% Cannabidiol cream (AVCN583601) for 4 weeks.

Full study procedures (phase II of the trial), see below:

Visit 1: Screening Visit: A screening form will be completed and patients who are willing to enroll and meet the eligibility criteria will be asked to sign the consent/assent form . Patients already on cannabinoids will be instructed to discontinue their treatment two weeks prior to the next visit (wash-out period). Subjects who were not treated with antibiotics or corticosteroids in the previous 2 weeks for topical and 4 weeks for systemic agents will start the trial at this time.

Visit 2: Baseline Visit: A baseline data collection form will be completed. We will select for the study treatment a chronic wound (present for more than 4 weeks), not measuring more than 1000 cm2. The surface area of the wound and quality of the wounds will be assessed and documented using the SWIFT medical wound assessment app, a validated tool that allows serial estimates and measurements of the wound surface areas. Bacterial swabs of selected target wound and medical photographs of the target wounds will be taken. For the pain intensity assessment, we will use a 100 mm visual analog scale (VAS), where 0 is no pain and 10- the worst pain ever experienced, while the DN4 scale will be used for assessment of neuropathic pain. For itch assessments, we will ask patients to determine the degree of itching experienced that day using a 100 mm horizontal VAS for itch. Patients will be provided with the study medication during this study visit and instructed to apply the cream twice a day for 4 weeks.

Blood sample (3 ml) will be taken to measure cannabinoid level in the blood. Visit 3: End of study visit: Patients will be assessed at 4 weeks when we will evaluate tolerability of the CBD oil and safety (e.g. burning sensation, pain, itch, local irritation, systemic symptoms). In addition, we will calculate the surface area change from previous visit as well as the characteristics of the wounds using the SWIFT medical wound assessment app. Patients will also be asked to score the average pain (VAS and DN4) and itching at the wound site for the prior 2 weeks and to complete a 100 mm VAS of wound change where -100 is the wound is double in size, 0- no change, and +100, wound is completely closed. Medical photographs of the target wounds will be taken.

Blood sample (3 ml) will be taken to measure cannabinoid level.

The study participants, completed phase II , who are willing to take part in phase III, will be able to participate , if eligible ( after appropriate wash out period).

Phase III will be a randomized, placebo controlled, blinded study ( Right versus Left side extremity), assessing the efficacy and safety CBD cream in EB patients with acute and chronic wounds.

30 EB patients with chronic or/and acute wounds, will participate in phase III. Randomization and Blinding: The name of each patient will be submitted to the research pharmacist. He will prepare a randomization scheme and will allocate patients' extremity to either placebo or CBD cream. Families and patients, as well as investigators will be blinded to the type of intervention throughout the duration of the study.

The intervention is CBD 3% cream / placebo. The study medications will be dispensed as 100 g jars. The study treatment will be applied to the entire or selected area of the extremity twice a day for 8 weeks (a drawing will be provided to the patients and to the assessors for the purpose of consistency).

The "placebo" will consist of a cream formulation with same color, consistency and smell as the intervention which will be applied on the other extremity (the application will mirror the process for the active medication).

Both jars will be labeled appropriately with the location and dosage instructions.

Allowable therapies: Patients will continue the same skin care routine and dressings with the exceptions of use of topical corticosteroids and topical antibiotics. Dressings that are impregnated with antimicrobials (silver, PHMB, honey, etc) are allowed if previously used.

Procedures: For the purpose of this phase we will select 2 different patient populations: A: acute wounds group (wounds that have been present for less than 4 weeks; B: chronic wounds group (wounds that have been present for >4 weeks) seen in patients with more severe types of EB.

For patients who have more than one chronic wound in the selected extremity we will add the individual wounds' surface areas.

Visit 1: Screening Visit: A screening form will be completed and patients who are willing to enroll and meet the inclusion criteria will be asked to sign the consent/assent form by our study nurse. Patients already on topical or systemic cannabinoids will be instructed to discontinue their treatment two weeks prior to the next visit (Wash-out period).

Visit 2: Baseline Visit:

In addition to the demographic and clinical, disease specific characteristics we will collect the following data:

Blister count, open and closed wound count, evidence of infection, dyspigmentation, EB nevi.

For patients with chronic wounds: surface area, wound characteristics , wound swab for culture and sensitivity, Current wound care regimen Pain score (VAS and DN4) Itch score iscorEB (clinician and patient) EBQOL CBD level (blood sample 3 ml)

Visit 3: Mid study visit (4 weeks): We will collect the same information as for baseline visit (Visit 2) and additional data:

VAS improvement patient Adverse events

Visit 4: End of study visit (8 weeks): We will collect the same information as for previous visit (Visit 3) , plus - the CBD level in the blood will be measured again ( 3 ml sample).

Wound swab will be taken ( group B), if the study investigator deems it is necessary.

ELIGIBILITY:
Inclusion Criteria:(phase 2) Patients 4-50 years of age

* Diagnosis of RDEB (clinically and/or molecular diagnosis)-
* Wounds that have not been healing for over 4 weeks
* Signed consent/assent form Inclusion criteria -Phase 3
* Patients 4-50 years of age
* Diagnosis of EB (clinically and/or molecular diagnosis)
* Evidence of either acute or chronic wounds on both extremities
* Patients enrolled in phase II are also eligible for participation in this phase, if they meet the current criteria and are interested in participation * Signed consent/assent form

Exclusion Criteria:

* Previous known allergy or intolerance to CBD cream

  * Topical and systemic use of cannabinoids in the past 2 weeks
  * Topical use of antibiotics, corticosteroids for the past 2 weeks
  * Other systemic medications that will interfere with the wound healing (corticosteroids, immunosuppressives, antibiotics) in the past 4 weeks
  * Surgery of the selected area in the past 8 weeks
  * Patients received medications metabolized via CYP3A4 enzyme (ketoconazole, itraconazole, ritonavir, clarithromycin, phenobarbital, rifampicin, carbamazepine, hexobarbital) for the past 2 weeks
  * Pregnancy

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Group A (patients with acute wounds). Difference in the total wound count (blister, open and closed wounds) compared to baseline | 8 weeks
  Difference in the total wound count (blister, open and closed wounds) compared to baseline
Group B (patients with chronic wounds). Percent change in the surface area of patients treated vs patients on placebo compared to baseline | 8 weeks
  Percent change in the surface area of patients treated with CBD vs patients on placebo compared to baseline
Group B (patients with chronic wounds). Proportion of treated patients that had more than 75% wound shrinkage | 8 weeks
  Proportion of patients that had more than 75% wound shrinkage (on the side of the body treated with CBD - in phase 3), compared to baseline.
Group B. Proportion of treated patients that had more than 50% wound shrinkage | 8 weeks
  Proportion of patients that had more than 50% wound shrinkage (on the side of the body treated with CBD - in phase 3), compared to baseline.
Percent changes in pain scores compared to baseline | 8 weeks
  Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (0 -no pain) and on the right (10- worst pain ever). The patient is asked to mark their pain level on the line at each study visit. The pain is scored using the VAS by measuring the distance in centimeters (0-10) from the "no pain" anchoring point.
  Difference in the pain score assessed using VAS, reported by the patient, between baseline and week 4, and week 8 visits will be calculated and multiplied by 10 to get result in percents(%).
Percent changes in itch scores compared to baseline | 8 weeks
  The intensity of itch is measured using the Visual Analog Scale for itch (VAS).It is a 10 cm line with anchor statements on the left (0- no itching) and on the right (10 -worst possible itching). The patient is asked to mark the intensity of itch on the line at each study visit. The itch is scored using the VAS by measuring the distance in centimeters (0-10) from the "no itch" anchoring point. the difference in the itch score as assessed using VAS( reported by the patient) between the first and visits Week 4 and Week 8, will be multiplied by 10 to get result in percents.
Percent changes in iscorEB (instrument for scoring clinical outcomes for research of EB), patient and clinician scores compared to baseline | 8 weeks
  iscorEB is a measurement tool for evaluating the disease severity in EB patient. It evaluates the cutaneous, mucosal and other organ impact of EB and includes clinician and patient reported outcomes in a single instrument. Score ranges between 0-120 for both reported outcomes. Patient portion of this instrument contains 15 questions. Each question has a score range from 0-8.Total score range for iscorEB patient portion is between 0 and 120. Reduction in iscorEB scores indicates improvement. An increase in score indicates deterioration. The difference in total patient and clinician scores between baseline and Week 4 ,8 visits will be divided by 120 ( max score for each portion)and multiplied by 100, to get the results in percents.
Percent changes in Quality of Life in Epidermolysis Bullosa Questionnaire score (QOLEB) EBQOL scores compared to baseline | 8 weeks
  QOLEB is a measurement tool containing 17 questions. Each question has a score range from 0-3.Total score range is between 0 and 51.
  Difference in the total scores between baseline and the study visits week 4, 8, will be divided by 51 and multiplied by 100 to get the result in percents.
correlation between patient's impression of improvement (VAS) and objective tools | 8 weeks
  Patient's impression of improvement is measured using the Visual Analog Scale (VAS).
  It is a 10 cm line with 3 anchor statements: on the left -"worsening", mid- "no changes", and on the right - "improvement". The patient is asked to mark his/her impression of improvement on the line at the final study visit. It will be scored by measuring the distance in centimeters (0-5) from the "no changes" anchoring point. The difference in this score as assessed using VAS( reported by the patient) between the baseline and EOS visit ,will be multiplied by 20 to get result in percents.

SECONDARY OUTCOMES:
• Percentage of patients that needed to stop the medication as a result of an adverse event | 8 weeks
  • Percentage of patients that needed to stop the medication as a result of an adverse event
Percentage of patients who experienced a serious adverse event | 8 weeks
  Percentage of patients who experienced a serious adverse event
Percentage of patients who had detectable levels of CBD in the blood | 8 weeks
  Percentage of patients who had detectable levels of CBD in the blood at the end of study visit.
• Percentage of patients who had clinical and laboratory evidence of infection in the wounds | 8 weeks
  • Percentage of patients who had clinical and laboratory evidence of infection in the wounds

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No